CLINICAL TRIAL: NCT03508674
Title: Prospective Study of Liver Mobilization With the Levita Magnetic Surgical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP003
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Levita Magnetic Surgical System
  Interventions: Device: Levita Magnetic Surgical System

INTERVENTIONS:
Device: Levita Magnetic Surgical System — use of surgical tool

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Levita Magnetic Surgical System in patients undergoing bariatric procedures

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm, open label study designed to assess the safety and effectiveness of the Levita Magnetic Surgical System in bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* scheduled to undergo bariatric procedure

Exclusion Criteria:

* Am Soc Anesthesiology score of III or IV
* significant comorbidities
* subjects contraindicated for use of magnetic system
* clinical history of impaired coagulation
* hepatic abnormality or anatomical abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Portenier, MD, Principal Investigator — Duke Regional Hospital
Locations (1):
- Hospital La Florida, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luengas R, Galindo J, Castro M, Marambio A, Watkins G, Rodriguez Del Rey M, Davanzo C, Portenier D, Guerron AD. First prospective clinical trial of reduced incision bariatric procedures using magnetic liver retraction. Surg Obes Relat Dis. 2021 Jan;17(1):147-152. doi: 10.1016/j.soard.2020.08.017. Epub 2020 Aug 26. PMID 33011073

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 54
Completed | 50
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 54

OUTCOME MEASURES:

1. Primary Outcome: Number and Types of Additional Tools Required to Mobilize the Liver During Procedure
Description: The ability to mobilize the liver will be evaluated by recording the number and types of additional tools used to mobilize the liver during a bariatric procedure. If another tool besides the Magnetic Surgical System (MSS) is required to move the liver then the use of the MSS has not been successful.
Time Frame: During planned bariatric procedure. (approximately 2 hours on a single day.)
Measure: Number; unit: Additional Tools to Mobilize Liver
Arm/Group | Intervention
Number analyzed (Participants) | 54
Additional Tools to Mobilize Liver | 0

2. Primary Outcome: Number of Participants With Adverse Events and Device Related Adverse Events
Description: All adverse events will be recorded and allocated as to relatedness to device, procedure or other.
Time Frame: Through 30 days post bariatric procedure
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 54
participants
  Total Participants With Adverse Events | 17
  Participants With Adverse Events Related to Device | 14

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 2/54
Other Adverse Events (participants affected / at risk) | 15/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=54)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abdominal Pain and Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=54)
Petechiae (Skin and subcutaneous tissue disorders) | 8 (8)
Liver Capsule Superficial Erosion Without Bleeding (Hepatobiliary disorders) | 7 (7)
Liver Capsule Superficial Abrasion Without Bleeding (Hepatobiliary disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hepatic Hematoma (Hepatobiliary disorders) | 1 (1)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT03508674/Prot_SAP_000.pdf